CLINICAL TRIAL: NCT04576741
Title: Testing the Feasibility and Acceptability of a Blended Mindfulness-Based Intervention for Persistent Depression
Brief Title: Blended Mindfulness-Based Intervention for Persistent Depression
Acronym: bMBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Mind and Life Europe (Unknown); Surrey and Borders Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPON/2020/08/FHMS
Record Dates: First submitted 2020-09-01; First posted 2020-10-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Persistent Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bMBI standard practice (Experimental): This is a 12-week online mindfulness-based course blended with therapist support via video link using standard practices for Mindfulness-Based Cognitive Therapy (30-minutes/day).
  Interventions: Behavioral: bMBI standard practice
- bMBI shorter more frequent practice (Experimental): This is a 12-week online mindfulness-based course blended with therapist support via video link using shorter, more frequent practice than standard Mindfulness-Based Cognitive Therapy (2x15-minutes/day).
  Interventions: Behavioral: bMBI shorter more frequent practice

INTERVENTIONS:
Behavioral: bMBI standard practice — This is a 12-week online mindfulness-based course blended with therapist support via video link using standard practices for Mindfulness-Based Cognitive Therapy (30-minutes/day).
  Arms: bMBI standard practice
Behavioral: bMBI shorter more frequent practice — This is a 12-week online mindfulness-based course blended with therapist support via video link using shorter, more frequent practice than standard Mindfulness-Based Cognitive Therapy (2x15-minutes/day).
  Arms: bMBI shorter more frequent practice

SUMMARY:
We plan to share all IPD but not any personal information.

ELIGIBILITY:
Inclusion criteria:

1. A current diagnosis of Major Depression as assessed by Structured Clinical Interview for DSM IV (First, Spitzer, Gibbon, & Williams, 2002).
2. A chronic or recurrent lifetime history of depression, with either chronic persistence of symptoms or a history of at least three previous episodes of depression, two of which needed to have occurred during the last two years.
3. Self-reported severity of current symptoms on a clinical level as indicated by a PHQ-9 score of 10 or more.
4. Age 18 to 65 thus excluding cases of late life depression given that such cases might diﬀer in aetiology.
5. Fluency in spoken and written English.
6. Have individual access to a computer or mobile device with internet connection and video link.

Exclusion criteria:

1. History of schizophrenia, schizoaffective disorder, bipolar disorder, current abuse of alcohol or other substances, organic mental disorder, pervasive developmental delay, primary diagnosis of obsessive-compulsive disorder or eating disorder, or regular nonsuicidal self-injury.
2. Current treatment with CBT more than once a month.
3. Regular meditation practice (meditating more than once per week).
4. Inability to complete research assessments through difficulty with English, visual impairment, or cognitive difficulties.
5. We will allow patients who are currently taking antidepressants into the study provided that the medication has not been changed during the last four weeks before entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Reductions in depression symptomatology as assessed using the Patient Health Questionnaire-9 (PHQ-9), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The PHQ-9 has 9 questions to assess the presence and severity of depression according to DSM-IV criteria and takes less than 3 minutes to complete. The PHQ-9 asks about patients' experiences in the last 2 weeks in relation to depression. Responses range from "0" (not at all) to "3" (nearly every day). Presence and severity of depression is scored as follows: 0-4 = minimal, 5-9 = mild, 10-14 = moderate, 15-19 moderately severe, 20-27 = severe.
  The PHQ-9 has been found to have a high level of validity and reliability (Kroenke, Spitzer, & Williams, 2001).

SECONDARY OUTCOMES:
Ability to decenter as assessed by self-report on the Experiences Questionnaire (EQ), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The EQ is a questionnaire to assess the ability to decenter. Decentering is defined as 'the ability to observe one's thoughts and feelings as temporary, objective events in the mind, as opposed to reflections of the self that are necessarily true' (Fresco et al., 2007). Decentering is thought to be a key mechanism for mindfulness-based interventions (Bernstein et al., 2019). There are 20 items and responses are made on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). We expect to see an increase in patient's ability to decenter.
  Convergent and discriminant validity has been shown in negative relationships with measures of depression symptoms, depressive rumination, experiential avoidance, and emotion regulation. Results have been replicated in clinical and non-clinical populations (Fresco et al., 2007).
Levels of mindfulness in daily life as assessed using the Five-Facet Mindfulness Questionnaire (FFMQ-15), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The FFMQ-15 is a questionnaire to assess levels of mindfulness in daily life. It assesses five aspects (or facets) of mindfulness: observation (noticing our internal and external environment), description (verbally labelling our experiences), mindful actions (acting with awareness), non-judgmental (not being overly critical of ourselves and others) and non-reactivity (not reacting impulsively to thoughts and feelings). The FFMQ-15 is the short version and has 15 items, the original version has 39. Responses are made on a 5-point Likert scale and range from 1 (never or rarely true) to 5 (very often or always true). There is a combination of direct scoring (e.g. 5=5) and reverse scoring (e.g. 5=1) to reveal a score for each facet and an overall total.
  The FFMQ-15 has been found to have high validity and reliability (Baer et al., 2006; Bohlmeijer et al., 2011).
Mind wandering and spontaneous thoughts as assessed by the Amsterdam Resting-State Questionnaire 2.0 (ARSQ 2.0), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The ARSQ 2.0 is a questionnaire to assess patients' subjective experience of their thoughts and feelings at rest. The questions tap into 10-factors: Discontinuity of Mind, Theory of Mind, Self, Planning, Sleepiness, Comfort, Somatic Awareness, Health Concern, Visual Thought and Verbal Thought. The ARSQ 2.0 involves a 5-minute eyes closed rest period followed by 55 questions about thoughts and feeling that were experienced. Responses are made on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). We expect to see an increase in Comfort and a decrease in Discontinuity of Mind.
  The test-retest correlations were found to be high for all 10-factors and mental health positively correlated with Comfort and negatively with Discontinuity of Mind (Diaz et al., 2013; Diaz et al., 2014).
Symptoms of anxiety as assessed using the Generalised Anxiety Disorder Assessment (GAD-7), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The GAD-7 is a questionnaire to assess the presence and severity of generalized anxiety disorder (GAD). It asks about patients' experiences in the last 2 weeks in relation to anxiety. Responses range from "0" (Not at all) to "3" (nearly every day). Presence and severity of anxiety is scored as follows: 0-5 = mild, 6-10 = moderate, 11-15 = moderately severe, 15-21 severe.
  The GAD-7 has been found to have good reliability, as well as criterion, construct, factorial, and procedural validity (sensitivity 89% and specificity 82%). Although anxiety and depression are closely related, factor analysis confirmed them as distinct dimensions. Also, good agreement was found between self-report and interviewer administered versions of the scale (Spitzer, Kroenke, Williams, & Loewe, 2006).
Subjective levels of stress as assessed using the Perceived Stress Scale (PSS), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The PSS is measure of the perception of stress and measures the degree to which situations in one's life are appraised as stressful. It is one of the most widely used measures of stress. There are 10 items that tap into how unpredictable, uncontrollable, and overloaded respondents find their lives. Questions ask about feelings and thoughts during the last month in relation to stress, enquiring how often they felt a certain way. Responses range from "0" (never) to "4" (very often). Scores are then reversed and summed to reveal at total between 0 and 40. Presence and severity of stress is scored as follows: 0-13 = low, 14-26 = moderate, 27-40 = high.
  The PSS has been found to have a good level of validity and reliability. (Cohen, Karmack, & Mermelstein, 1988; Roberti et al., 2006; Taylor, 2015).
Mental wellbeing as assessed using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), change measured within 1 week of starting and finishing the course and in week 5 and 9. | Weeks 0, 5, 9,13.
  The WEMWBS is a measure of mental wellbeing. There are 14 items that enquire about both the feeling (e.g. I have been feeling cheerful) and functioning (e.g. I have been feeling useful) aspect of mental wellbeing. Responses range from "0" (none of the time) to "5" (all of the time). Scores are summed to reveal a total between 14 and 70. Based on UK population samples: 14-42 = low wellbeing, 43-59 = average wellbeing, 60-70 = high wellbeing.
  The WEMWBS has been used extensively worldwide and has been found to have high validity and reliability (Clarke et al., 2011; Taggart et al., 2013; Maheswaran at al., 2012).

OTHER OUTCOMES:
Levels of engagement assessed by participants filling out a simple form each day to record which activities they have completed that day. | Daily from weeks 1 to 12.
  Participants will fill out a simple form at the end of each day to record which activities they have been able to complete. This will allow us to assess levels of engagement in the intervention and how this is correlated with clinical outcomes.
Practice adherence and skills utilization will be assessed by participants replying to several short messages each day sent to their mobile phone. | Daily from weeks 1 to 12.
  Effects on practice adherence and skills utilization will be investigated using experience sampling methodology (a method of recording subjective experiences in daily life). Participants will respond to several short messages a day sent to their mobile phone about their daily subjective experiences. This will allow us to assess patients in the moment subjective experience rather than their retrospective subjective experience.
Participants' views on acceptability, barriers and facilitators to engagement, and their experience and utilization of mindfulness skills, will be assessed in a post-intervention interview via video link, within 1 week of finishing the course. | Week 13.
  Qualitative assessments will be conducted during a post-intervention interview via video link. They will serve to assess patients' views on acceptability of the intervention and practices, their experience and utilization of mindfulness skills, and their views on potential barriers and facilitators of engagement. Qualitative assessments will be based on a semi-structured topic guide. The interview will last about 30 minutes. Interviews will be transcribed and subjected to thematic analysis using a framework approach.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hamilton, Principal Investigator — University of Surrey
Locations (1):
- Surrey and Borders Partnership NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes